CLINICAL TRIAL: NCT00230724
Title: Maintaining Exercise After Cardiac Rehabilitation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: HL76734
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2005-10-03 (Estimated); Status verified 2005-09

CONDITIONS: Cardiovascular Disease
Keywords: Exercise maintenance
MeSH Terms: conditions — Cardiovascular Diseases

INTERVENTIONS:
Behavioral: Exercise Counseling

SUMMARY:
Maintaining exercise participation among patients who have completed cardiac rehabilitation is integral to secondary prevention of coronary events and cardiac re-hospitalization. To promote exercise maintenance after completion of a 12 week Phase II rehabilitation program, we propose to offer a theoretically-based intervention that we have used successfully to promote exercise among older, primary-care patients. This program (Maintenance Counseling) includes brief advice from the Cardiac Rehabilitation case manager at Phase II program discharge followed by telephone-counseling based on the Transtheoretical Model of Behavior Change and Social Cognitive Theory. Health educators will provide the telephone-based intervention over 6 months. Using a randomized controlled design, 180 patients will be assigned to Maintenance Counseling or Brief Advice plus Contact Control. Outcome assessments will include an exercise tolerance test (baseline/post-rehabilitation and 6 months), self-reported exercise participation, motivational readiness for exercise, and objective activity monitoring at baseline, 6, 12 and 18 months.

DETAILED DESCRIPTION:
Maintaining exercise participation among patients who have completed cardiac rehabilitation is integral to secondary prevention of coronary events and cardiac re-hospitalization. Patients in Phase II cardiac rehabilitation programs, a majority being older adults, participate in regular supervised exercise during the program; however, long-term adherence to exercise is poor, with only 30% reporting regular exercise at 12 month follow-ups. To promote exercise maintenance after completion of a 12 week Phase II rehabilitation program, we propose to offer a theoretically-based intervention that we have used successfully to promote exercise among older, primary-care patients. This program (Maintenance Counseling) includes brief advice from the Cardiac Rehabilitation case manager at Phase II program discharge followed by telephone-counseling based on the Transtheoretical Model of Behavior Change and Social Cognitive Theory. Health educators will provide the telephone-based intervention over 6 months. Using a randomized controlled design, 180 patients will be assigned to Maintenance Counseling or Brief Advice plus Contact Control. Outcome assessments will include an exercise tolerance test (baseline/post-rehabilitation and 6 months), self-reported exercise participation, motivational readiness for exercise, and objective activity monitoring at baseline, 6, 12 and 18 months. These data will help to identify whether telephone-based exercise counseling is an effective strategy for sustaining regular exercise and fitness among cardiac rehabilitation patients thereby contributing to secondary prevention of coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:: 1) men and women aged >40 years participating in supervised Phase II CR. The CR population tends to be older (mean age: 64.5+11.9, range 38-83 years, Preliminary Studies C.6.) and by including adults as young as 40 years, we expect to offer the program to the majority of Phase II CR patients. (2) scheduled to complete Phase II CR in the next 4 weeks, 3) able to read and speak English, 4) provide consent for medical chart review to extract disease and treatment variables, 5) able to walk unassisted. 6) We plan to include patients who participated in Phase II CR due to a diagnosis of coronary heart disease (e.g., post- MI, CABG, chronic angina pectoris) or chronic heart failure.

-

Exclusion Criteria:1) Prior neurological brain disorder (e.g., Seizure Disorder, Traumatic Brain Injury. Patients with prior neurological disease, including large vessel stroke and Alzheimer's Disease will be excluded. 2) An arbitrary Mini-Mental Status Examination (MMSE) cutoff score of >10 will be set to exclude patients whose scores suggest dementia or cognitive impairments that will interfere with ability to provide informed consent and complete research demands.

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2005-04; Study Completion 2007-04

PRIMARY OUTCOMES:
Participation in exercise (weekly minutes of exercise) at 6 months.

SECONDARY OUTCOMES:
Fitness on a sub-maximal graded stress test
Weekly minutes of exercise at 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernardine M Pinto, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- Center for Cardiac Fitness, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Pinto BM, Dunsiger SI. Mediators of exercise maintenance after cardiac rehabilitation. J Cardiopulm Rehabil Prev. 2015 Jan-Feb;35(1):13-20. doi: 10.1097/HCR.0000000000000065. PMID 24983707
- [Derived] Pinto BM, Goldstein MG, Papandonatos GD, Farrell N, Tilkemeier P, Marcus BH, Todaro JF. Maintenance of exercise after phase II cardiac rehabilitation: a randomized controlled trial. Am J Prev Med. 2011 Sep;41(3):274-83. doi: 10.1016/j.amepre.2011.04.015. PMID 21855741